CLINICAL TRIAL: NCT06692855
Title: Prognostic Value of the Rockwood Clinical Frailty Score in Cardiogenic Shock
Acronym: FrailShock
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9454
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Cardiogenic Shock
Keywords: Cardiogenic shock; CardShock risk score; Area under the curve (AUC); SCAI Shock classification; Clinical Frailty Scale (CFS)
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiogenic shock (CS) is characterized by tissue hypoperfusion resulting from cardiac dysfunction, without hypovolemia, where the ventricular pump is unable to generate adequate blood flow to meet the metabolic needs of the organs.

To date, the management of CS is a challenge for cardiologists and intensive care physicians, particularly with regard to the stratification of the severity of these patients to accurately determine the prognostic outcome. Thus, although specific prognostic scores for CS already exist, they are often inefficient and difficult to calculate quickly at the patient's bedside. For example, the CardShock risk score is a score composed of seven variables (including biological and echocardiographic parameters) allowing in the best case to obtain an area under the curve (AUC) for the prediction of mortality around 0.7. More recently, the SCAI Shock classification was developed to progressively stratify patients into five groups of increasing severity, ranging from A to E for the most serious. Although its prognostic interest is better than the CardShock, this recently updated classification is also based on biological or echocardiographic parameters that are sometimes difficult to collect in an emergency.

Thus, there is currently no simple and optimal prognostic score to predict the prognosis of patients and even less of a score that takes into account the overall clinical fragility of patients appropriately.

In this context, the Rockwood clinical fragility score, also called the "Clinical Frailty Scale" (CFS), has emerged in recent years as an iconographic score accompanied by an explanatory text initially developed to assess fragility in the elderly. It is a pure declarative score, very easy to perform in clinical practice, even in acute situations or in delirious or even sedated patients. It also has the advantage of being free since it only groups together the physiological and functional data characterizing the previous state of a subject before the diagnostic and therapeutic stage. The CFS makes it possible to estimate the degree of fragility of a patient ranging from "very fit" or robust, active, energetic to "terminal phase". It is based on information that is easily retrieved from the patient or the patient's relatives with the advantage of having a very good correlation with the fragility scores that are more complex to evaluate.

Finally, the CSF has already proven its worth in acute cardiology, such as in myocardial infarction where this score was independently and strongly associated with all-cause mortality at 6 months and where it was highlighted that fragile patients had a poorer outcome, a higher risk of mortality, risk of CS and risk of bleeding.

Optimal management of CS patients requires both a thorough, rapid, reliable and easy-to-obtain assessment in an emergency in order to initiate appropriate interventions as quickly as possible. In this perspective, the CFS emerges as a promising parameter in the initial assessment of these patients, particularly to identify patients with a higher risk of complications. This score alone or in addition to the scores already used in practice in the CS represents an innovative perspective and could allow a more detailed assessment of patients and thus help clinicians to better target the necessary interventions and to individualize the management. Indeed, optimizing the identification of patients with acute critical cardiology is one of the avenues suggested as an area for improvement by experts in this field at the border of cardiology and resuscitation. The simplicity of this tool, combined with its ability to assess the overall vulnerability of the patient, opens the way to increased personalization of care in CS patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18 years)
* Patient with cardiogenic shock according to ESC 2021 definition
* Patient hospitalized from January 1, 2014 to September 1, 2024 in an Intensive Care Unit
* Patients who do not object to the re-use of their data for the purposes of this research.

Criteria Exclusion:

* Patient having expressed his opposition to the re-use of his data for scientific research purposes.
* Subject under court protection.
* Subject under guardianship or curatorship.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patient (≥18 years) with cardiogenic shock according to ESC 2021 definition
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Death at 28 days after cardiogenic shock | 28 days after cardiogenic shock

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Médecine Intensive - Réanimation - CHU de Strasbourg - France, Strasbourg, France